CLINICAL TRIAL: NCT04615195
Title: Effect of COVID-19 Related COntainment in ChildreN
Acronym: E-COCCON
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0205
Record Dates: First submitted 2020-11-03; First posted 2020-11-04 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children between 8 and 15 years old: answer to the CRIES 13 questionnaire
  Interventions: Other: cries 13 questionnaire

INTERVENTIONS:
Other: cries 13 questionnaire — Participant will be contacted by telephone by a clinical research assistant to answer the CRIES 13 questionnaire.
  In large families, the CRIES-13 of the holder of parental authority and of the child will be applied for each of them whose age corresponds to the inclusion criteria.

SUMMARY:
The current pandemic situation (SRAS COV2) is an unprecedented event and a source of stress potentially aggravated by containment. The Child Revised Impact Event Scale (CRIES-13) was evaluated in children 8 years or older in survivors of traumatic events, flood, stay in intensive care, or war (Bosnia). In this study CRIES-13 will be used to determine the prevalence of precursor signs of post-traumatic stress in children aged 8 to 15 confined between March 17, 2020 and May 2020

DETAILED DESCRIPTION:
Parents of children aged 8 to 15 will be approached from different levels / places of selection / recruitment. A clinical researcher of pediatric clinical investigation center will collect the responses.

If one of the holders of parental authority and the child agree to participate, an information notice will be sent to them, then they will be contacted by telephone by a clinical research assistant to answer the questionnaire.

In large families, the CRIES-13 of the holder of parental authority and of the child will be applied for each of them whose age corresponds to the inclusion criteria.

The duration of the study / participant call and effective response to the questionnaire by the holder of parental authority and the child will takes a maximum of 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Binomial of child (aged between 8 and 15) and one of its holders of parental authority agreeing to participate

Exclusion Criteria:

* children aged under 8 and over 15
* children whose parents are opposed
* children refusing to participate
* holders of minor parental authority

Ages: 8 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: All children aged between 8 and 15 accepting to participate and whose parents accepting to particpate
Sampling Method: Non-Probability Sample
Enrollment: 703 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Signs of post traumatic stress disorder | 1 month
  Using a simple score (Child Revised Impact of Event Scale (CRIES-13)), determine the prevalence of precursor signs of post-traumatic stress in children aged 8 to 15 confined between March 17, 2020 and May 2020

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Claudet, Pr, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Claudet I, Marchand-Tonel C, Ricco L, Houze-Cerfon CH, Lang T, Brehin C. During the COVID-19 Quarantine, Home Has Been More Harmful Than the Virus for Children! Pediatr Emerg Care. 2020 Sep;36(9):e538-e540. doi: 10.1097/PEC.0000000000002205. No abstract available. PMID 32868552
- [Result] Claudet I, Marchand-Tonel C, Kelly-Irving M, Gaudron CZ, Raynaud JP, Delpierre C, Brehin C. The psychological effects of COVID-19-related containment in children: The E-COCCON French study. Arch Pediatr. 2022 Apr;29(3):188-193. doi: 10.1016/j.arcped.2022.01.011. Epub 2022 Jan 19. PMID 35115219